CLINICAL TRIAL: NCT04160975
Title: Persuasion in Medicine: Experimental Evidence on Sender and Signal Effects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard University (Other)
Collaborators: Ludwig-Maximilians - University of Munich (Other); Massachusetts Institute of Technology (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Marcella Alsan, Principal Investigator, Harvard University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: IRB19-1424
Record Dates: First submitted 2019-11-08; First posted 2019-11-13 (Actual); Results first posted 2021-06-29 (Actual); Last update posted 2021-06-29 (Actual); Status verified 2021-06

CONDITIONS: Flu, Human; Influenza, Human; Covid19
Keywords: Belief Updating; Preventive Care; Racial Disparity
MeSH Terms: conditions — Influenza, Human; COVID-19

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Black R/Race C/Doctor/Standard Script (Experimental): Video which contains a racially concordant actor playing a doctor and reading a standard script. The receiver of the message will be Black.
  Interventions: Behavioral: Video about safety and effectiveness of adult seasonal flu vaccination
- Black R/Race C/Layperson/Standard Script (Experimental): Video which contains a racially concordant actor playing a layperson and reading a standard script. The receiver of the message will be Black.
  Interventions: Behavioral: Video about safety and effectiveness of adult seasonal flu vaccination
- Black R/Race D/Doctor/Standard Script (Experimental): Video which contains a racially discordant actor playing a doctor and reading a standard script. The receiver of the message will be Black.
  Interventions: Behavioral: Video about safety and effectiveness of adult seasonal flu vaccination
- Black R/Race D/Doctor/Acknowledgement Script (Experimental): Video which contains a racially discordant actor playing a doctor and reading an acknowledgement script. The receiver of the message will be Black.
  Interventions: Behavioral: Video about safety and effectiveness of adult seasonal flu vaccination
- White R/Race C/Doctor/Standard Script (Experimental): Video which contains a racially concordant actor playing a doctor and reading a standard script. The receiver of the message will be White.
  Interventions: Behavioral: Video about safety and effectiveness of adult seasonal flu vaccination
- White R/Race D/Doctor/Standard Script (Experimental): Video which contains a racially discordant actor playing a doctor and reading a standard script. The receiver of the message will be White.
  Interventions: Behavioral: Video about safety and effectiveness of adult seasonal flu vaccination

INTERVENTIONS:
Behavioral: Video about safety and effectiveness of adult seasonal flu vaccination — The investigators will show subjects videos of either Black or white male actors providing scripted information on the flu vaccination. The content of the video will be the safety and effectiveness of adult seasonal flu vaccination. The videos contain one of Black or white actors playing the role of either a doctor or a layperson as well as different scripts.

SUMMARY:
The aim of the study is to identify what sender/signal combinations are most persuasive in encouraging low socioeconomic males living in the U.S. to take-up seasonal flu vaccination. The investigators plan to recruit male subjects and randomly assign them to four persuasion treatments: three of which vary dimensions of the sender of a medical recommendation (racial concordance and authority treatments) and one which varies the signal (standard vs. empathetic). Specifically, the investigators will show subjects videos of either Black or white actors/actresses providing scripted information on the flu vaccination. The investigators will randomize the race of the sender and if the subject is Black, also randomize the authority of the sender, with the actor portraying either a doctor or a layperson. In addition, the investigators will vary the script used in the experiment between one that acknowledges past injustices (indicated as an empathetic script hereafter) and one that does not (indicated as a standard script hereafter). The investigators will provide subjects a free flu shot coupon and elicit the price at which subjects would be willing to give up this coupon for a cash reward. Lastly, in light of the relevance of vaccination take-up in combating COVID-19 pandemic, the investigators will assess demand for information about a COVID-19 vaccine, with subjects invited to receive results of a safety and efficacy review from a trusted or standard source. The design requires the collection of baseline and endline surveys combined with administrative data from pharmacies about coupon redemption. The primary outcomes of interest are posterior beliefs about seasonal flu vaccination, demand and willingness-to-pay (WTP) for a free flu shot coupon, redemption of the coupon, and demand for information about a COVID-19 vaccine.

DETAILED DESCRIPTION:
The investigators will recruit approximately 3350 African-American or Caucasian adult males with a high-school diploma or less. A pilot study, which ran during the 2019-20 flu season, recruited approximately 850 subjects, and a planned scale-up will recruit an additional 2500 subjects during the 2020-21 flu season. The investigators will oversample African American individuals, emphasizing low-income and minority men because these characteristics are correlated with lower relative take-up of flu vaccination. After informed consent is obtained, subjects will be asked about sociodemographic information (age, education, income and marital status), healthcare experience and past medical history, knowledge and beliefs about flu vaccination, and location of the nearest pharmacy. The investigators will then randomly assign the adult male subjects to videos which contain one of Black or white actors playing the role of either a doctor or a layperson as well as different scripts. The content of the infomercial will be the safety and effectiveness of adult seasonal flu vaccination. After the video, the investigators will obtain information on beliefs regarding vaccination, feedback on the video, attention to the video and willingness-to-pay for a flu shot coupon. The final baseline module will consist of a randomly assigned invitation to receive the results of an upcoming review of a COVID-19 vaccine, with subjects assigned to receive information from a trusted or standard source. The investigators will track flu coupon redemption, which is redeemable at most pharmacies nationwide.

ELIGIBILITY:
Inclusion Criteria:

* Age: See above.
* Education: Less than a college degree.
* Gender: Male.
* Race: Caucasian or African American.
* Miscellaneous: Has not received the flu shot in the current flu season yet.
* Miscellaneous: Has sound on his device turned on.

Exclusion Criteria:

* Fast survey-taking: subjects who are among the 5% fastest in terms of total time spent on survey within race and treatment group.
* Nonsense answers (those that do not have decipherable English) in the open text sections that suggest low effort.
* Inconsistent responses to questions (such as being willing to give up $10 to receive a flu coupon but not $1).
* Repeat survey takers as indicated by duplicate emails or IP addresses in survey data.

Ages: 18 Years to 51 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — The investigators will only recruit male subjects.
Enrollment: 3245 (Actual)
Dates: Start 2019-12-20 (Actual); Primary Completion 2021-02-19 (Actual); Study Completion 2021-02-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Harvard University, Cambridge, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Black Participant-Concordant Sender-Expert Sender-Standard Signal: Black participants who are assigned to a concordant-exper sender delivering a standard signal.
- Black Participant-Concordant Sender-Lay Sender-Standard Signal: Black participants who are assigned to a concordant-lay sender delivering a standard signal.
- Black Participant-Discordant Sender-Expert Sender-Standard Signal: Black participants who are assigned to a discordant-exper sender delivering a standard signal.
- Black Participant-Discordant Sender-Expert Sender-Acknowledgement Signal: Black participants who are assigned to a discordant-exper sender delivering a acknowledgement signal.
- White Participant-Concordant Sender-Expert Sender-Standard Signal: White participants who are assigned to a concordant-exper sender delivering a standard signal.
- White Participant-Discordant Sender-Expert Sender-Standard Signal: White participants who are assigned to a discordant-exper sender delivering a standard signal.
Period: Overall Study
Arm/Group | Black Participant-Concordant Sender-Expert Sender-Standard Signal | Black Participant-Concordant Sender-Lay Sender-Standard Signal | Black Participant-Discordant Sender-Expert Sender-Standard Signal | Black Participant-Discordant Sender-Expert Sender-Acknowledgement Signal | White Participant-Concordant Sender-Expert Sender-Standard Signal | White Participant-Discordant Sender-Expert Sender-Standard Signal
Started | 479 | 496 | 478 | 485 | 649 | 658
Completed | 415 | 430 | 417 | 410 | 614 | 607
Not Completed | 64 | 66 | 61 | 75 | 35 | 51

BASELINE CHARACTERISTICS:
Population: Participants who were eligible to participate in and completed the baseline survey.
Groups:
- Total: Total of all reporting groups
Arm/Group | Black Participant-Concordant Sender-Expert Sender-Standard Signal | Black Participant-Concordant Sender-Lay Sender-Standard Signal | Black Participant-Discordant Sender-Expert Sender-Standard Signal | Black Participant-Discordant Sender-Expert Sender-Acknowledgement Signal | White Participant-Concordant Sender-Expert Sender-Standard Signal | White Participant-Discordant Sender-Expert Sender-Standard Signal | Total
Number analyzed (Participants) | 415 | 430 | 417 | 410 | 614 | 607 | 2893
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.92048 (6.717987) | 35.53023 (6.219959) | 36.1247 (6.46877) | 35.90488 (6.857133) | 38.11401 (6.773668) | 38.16474 (6.760583) | 36.82613 (6.742281)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 415 | 430 | 417 | 410 | 614 | 607 | 2893
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 415 | 430 | 417 | 410 | 0 | 0 | 1672
  White | 0 | 0 | 0 | 0 | 614 | 607 | 1221
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 415 | 430 | 417 | 410 | 614 | 607 | 2893
High School [Count of Participants; unit: Participants]
  Completed | 359 | 380 | 374 | 355 | 554 | 533 | 2555
  Not completed | 56 | 50 | 43 | 55 | 60 | 74 | 338
Married [Count of Participants; unit: Participants] | 71 | 86 | 89 | 77 | 202 | 186 | 711
Insured [Count of Participants; unit: Participants] | 234 | 251 | 245 | 239 | 403 | 391 | 1763
Subjective Health Status [Mean (Standard Deviation); unit: units on a scale] — Subjective Health Status is measured on a 5-point Likert scale (where 1 is poor and 5 is excellent).
  units on a scale | 3.522892 (1.009056) | 3.751163 (1.003925) | 3.642686 (1.0069) | 3.653659 (1.056843) | 3.21987 (.992071) | 3.237232 (.9965605) | 3.468372 (1.030375)
Subjective Flu Shot Cost [Mean (Standard Deviation); unit: dollar] | 43.91588 (91.2157) | 42.74393 (85.77928) | 38.14388 (79.24301) | 33.8441 (72.69948) | 25.28546 (50.80593) | 25.02221 (48.44235) | 33.56405 (70.94346)
Has Primary Care Provider [Count of Participants; unit: Participants] | 189 | 178 | 192 | 171 | 321 | 323 | 1374
(Prior) Flu Vaccine Intent [Mean (Standard Deviation); unit: units on a scale] — Flu vaccine intent is measured on a scale of 0 (extremely unwilling) to 10 (extremely willing).
  units on a scale | 2.554217 (3.243176) | 2.786047 (3.324808) | 2.446043 (3.307566) | 2.485366 (3.147713) | 2.596091 (3.146201) | 2.52883 (3.237376) | 2.566886 (3.228842)
(Prior) Likelihood of Contracting Flu [Mean (Standard Deviation); unit: units on a scale] — Likelihood of contracting flu is measured on a scale of 0 (extremely unlikely) to 10 (extremely likely).
  units on a scale | 2.342169 (2.853683) | 2.072093 (2.791414) | 2.143885 (2.823905) | 2.304878 (2.86659) | 2.760586 (2.603112) | 2.912685 (2.701415) | 2.476668 (2.774967)

OUTCOME MEASURES:

1. Primary Outcome: Rating of Sender
Description: This is an inverse-covariance-weighted index comprised of responses to survey questions regarding:
  1. whether the respondent was interested in further medical advice from the given sender (measured as a binary outcome);
  2. whether the respondent trusted advice from the sender measured on a scale of 1 to 5;
  3. and whether the respondent's assessment of the sender's qualification to provide medical advice measured on a scale of 1 to 5.
  It is standardized to a mean of 0 and standard deviation of 1. Scores less than 0 indicate lower ratings of the sender rated by participants in Arm A (described in each arm/group description) compared to the rating rated by participants in Arm B (also described in each arm/group description). Scores greater than 0 indicate higher ratings of the sender by Arm A compared to by Arm B. For example, an index score of .18 indicates that participants in Arm A rate the sender 0.18 index (in standard deviation units) higher than those in Arm B.
Time Frame: This outcome was assessed during Baseline survey, which took approximately 20 minutes.
Population: Arms/Groups are combined as described in each arm/group description in order to test hypotheses prespecified in the analysis plan as well as to measure the effect of the given intervention on the outcome among the group of participants in Arm A compared to Arm B. The intervention and Arms A and B are described in each arm/group description.
Measure: Number (95% Confidence Interval); unit: index
Groups:
- Concordant (Arm A) vs. Discordant Expert Sender (Arm B) - Black Participants: This group combines the following arms to measure the effect of racial concordance between sender and receiver (i.e. intervention) among Black Participants:
  1. Black Participant-Concordant Sender-Expert Sender-Standard Signal (i.e. Arm A)
  2. Black Participant-Discordant Sender-Expert Sender-Standard Signal (i.e. Arm B)
  The arms are combined to test Hypothesis 1 prespecified in the analysis plan. The hypothesis tests how racial concordance between an expert sender and receiver affects the outcome among participants assigned to Arm A compared to those who are assigned to Arm B.
- Concordant (Arm A) vs. Discordant Expert Sender (Arm B) - White Participants: This group combines the following arms to measure the effect of racial concordance between sender and receiver (i.e. intervention) among White Participants:
  1. White Participant-Concordant Sender-Expert Sender-Standard Signal (i.e. Arm A)
  2. White Participant-Discordant Sender-Expert Sender-Standard Signal (i.e. Arm B)
  The arms are combined to test Hypothesis 1 prespecified in the analysis plan. The hypothesis tests how racial concordance between an expert sender and receiver affects the outcome among participants assigned to Arm A compared to those who are assigned to Arm B.
- Acknowledgement (Arm A) vs. Standard Signal (Arm B) - Black Participants: This group combines the following arms to measure the effect of an acknowledgement signal (i.e. intervention) among Black Participants:
  1. Black Participant-Discordant Sender-Expert Sender-Acknowledgement Signal (i.e. Arm A)
  2. Black Participant-Discordant Sender-Expert Sender-Standard Signal (i.e. Arm B)
  The arms are combined to test Hypothesis 4 prespecified in the analysis plan. The hypothesis tests how a signal that acknowledges past injustices affects the outcome among participants assigned to Arm A compared to those assigned to Arm B.
- Layperson Sender (Arm A) vs. Expert Sender (Arm B) - Black Participants: This group combines the following arms to measure the effect of a layperson sender (i.e. intervention) among Black Participants:
  1. Black Participant-Concordant Sender-Lay Sender-Standard Signal (i.e. Arm A)
  2. Black Participant-Concordant Sender-Expert Sender-Standard Signal (i.e. Arm B)
  The arms are combined to test Hypothesis 3 prespecified in the analysis plan. The hypothesis tests how a layperson sender affects the outcome among participants assigned to Arm A compared to those assigned to Arm B.
Arm/Group | Concordant (Arm A) vs. Discordant Expert Sender (Arm B) - Black Participants | Concordant (Arm A) vs. Discordant Expert Sender (Arm B) - White Participants | Acknowledgement (Arm A) vs. Standard Signal (Arm B) - Black Participants | Layperson Sender (Arm A) vs. Expert Sender (Arm B) - Black Participants
Number analyzed (Participants) | 832 | 430 | 827 | 845
index | .1828917 [.0506082 to .3151752] | -.0750636 [-.1870341 to .0369069] | .0997998 [-.0345829 to .2341826] | -.5397662 [-.6789624 to -.4005701]

2. Primary Outcome: Rating of Signal
Description: This is an inverse-covariance-weighted index comprised of responses to survey questions on:
  1. recommending the video to friends and family measured on a scale of 0 to 10;
  2. recommending the flu shot to friends and family measured on a scale of 0 to 10;
  3. and the respondent's assessment of the extent to which the information contained in the video was useful measured on a scale of 1 to 5.
  It is standardized to a mean of 0 and standard deviation of 1. An index score of 0 is equal to the mean. Scores less than 0 indicate lower ratings of the signal rated by participants in Arm A (described in each arm/group description) compared to the rating rated by participants in Arm B (also described in each arm/group description). Scores greater than 0 indicate higher ratings of the signal by Arm A compared to by Arm B. For example, an index score of 0.14 indicates that participants in Arm A rate the signal 0.14 index (in standard deviation units) higher than those in Arm B.
Time Frame: This outcome was assessed during Baseline survey, which took approximately 20 minutes.
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: index
Arm/Group | Concordant (Arm A) vs. Discordant Expert Sender (Arm B) - Black Participants | Concordant (Arm A) vs. Discordant Expert Sender (Arm B) - White Participants | Acknowledgement (Arm A) vs. Standard Signal (Arm B) - Black Participants | Layperson Sender (Arm A) vs. Expert Sender (Arm B) - Black Participants
Number analyzed (Participants) | 832 | 1221 | 827 | 845
index | .1387205 [.0003558 to .2770851] | -.0088105 [-.1199617 to .1023406] | .1423725 [.0062946 to .2784504] | -.0806321 [-.2126516 to .0513873]

3. Primary Outcome: Signal Content Recall
Description: This is an inverse-covariance-weighted index comprised of responses to survey questions on:
  1. whether age group for whom the flu vaccine is recommended (measured as a binary outcome); and
  2. whether the flu shot contains the flu virus (recall of information discussed in the video) (measured as a binary outcome).
  It is standardized to a mean of 0 and standard deviation of 1. An index score of 0 is equal to the mean. Scores less than 0 indicate lower level of recalling signal content among participants in Arm A (described in each arm/group description) compared to the level among participants in Arm B (also described in each arm/group description). Scores greater than 0 indicate a higher level of recalling signal content among participants in Arm A compared to those in Arm B. For example, an index score of 0.02 indicates that participants in Arm A recall signal content 0.02 index (in standard deviation units) higher than those in Arm B.
Time Frame: This outcome will be assessed during Baseline survey, which takes approximately 20 minutes.
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: index
Arm/Group | Concordant (Arm A) vs. Discordant Expert Sender (Arm B) - Black Participants | Concordant (Arm A) vs. Discordant Expert Sender (Arm B) - White Participants | Acknowledgement (Arm A) vs. Standard Signal (Arm B) - Black Participants | Layperson Sender (Arm A) vs. Expert Sender (Arm B) - Black Participants
Number analyzed (Participants) | 832 | 1221 | 827 | 845
index | -.0062555 [-.1415234 to .1290124] | .0193832 [-.0926014 to .1313679] | .0041984 [-.131372 to .1397687] | .1166304 [-.0149457 to .2482066]

4. Primary Outcome: Safety Beliefs
Description: This is an inverse-covariance-weighted index comprised of:
  1. the point belief on the likelihood to contract the flu from the flu shot measured by a Likert scale and rescaled to have a support of -1 to 1.
  2. the certainty measured with a balls and bins method and rescaled to have a support of -1 to 1.
  It is standardized to a mean of 0 and standard deviation of 1. An index score of 0 is equal to the mean. Scores less than 0 indicate a lower level of beliefs in the safety of flu vaccine among participants in Arm A (described in each arm/group description) compared to the level among participants in Arm B (also described in each arm/group description). Scores greater than 0 indicate a higher level of beliefs among participants in Arm A compared to those in Arm B. For example, an index score of -0.1 indicates that participants in Arm A hold such beliefs 0.1 index (in standard deviation units) lower than those in Arm B.
Time Frame: This outcome will be assessed during Baseline survey, which takes approximately 20 minutes.
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: index
Arm/Group | Concordant (Arm A) vs. Discordant Expert Sender (Arm B) - Black Participants | Concordant (Arm A) vs. Discordant Expert Sender (Arm B) - White Participants | Acknowledgement (Arm A) vs. Standard Signal (Arm B) - Black Participants | Layperson Sender (Arm A) vs. Expert Sender (Arm B) - Black Participants
Number analyzed (Participants) | 832 | 1221 | 827 | 845
index | -.0979564 [-.2331252 to .0372124] | -.027714 [-.1410194 to .0855914] | -.1065867 [-.2425802 to .0294069] | -.0242752 [-.1580924 to .109542]

5. Primary Outcome: Coupon Interest
Description: This is an inverse-covariance-weighted index comprised of revealed preference measures of demand for a free flu shot coupon:
  1. Willingness to pay (WTP) for the coupon measured as $0, $1, $2, $5, or $10
  2. demand for information regarding locations to redeem the coupon measured as a binary outcome
  It is standardized to a mean of 0 and standard deviation of 1. An index score of 0 is equal to the mean. Scores less than 0 indicate a lower level of interest in a free flu shot coupon distributed after survey completion among participants in Arm A (described in each arm/group description) compared to the level among participants in Arm B (also described in each arm/group description). Scores greater than 0 indicate a higher level of interest among participants in Arm A compared to those in Arm B. For example, an index score of -0.01 indicates that participants in Arm A hold such interest -0.01 index (in standard deviation units) higher than those in Arm B.
Time Frame: This outcome was assessed during Baseline survey, which took approximately 20 minutes.
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: index
Arm/Group | Concordant (Arm A) vs. Discordant Expert Sender (Arm B) - Black Participants | Concordant (Arm A) vs. Discordant Expert Sender (Arm B) - White Participants | Acknowledgement (Arm A) vs. Standard Signal (Arm B) - Black Participants | Layperson Sender (Arm A) vs. Expert Sender (Arm B) - Black Participants
Number analyzed (Participants) | 832 | 1221 | 827 | 845
index | -.0078177 [-.1389825 to .123347] | -.0827849 [-.1924382 to .0268684] | .0280955 [-.1069421 to .1631332] | -.0162865 [-.1513941 to .1188211]

6. Primary Outcome: (Posterior) Flu Vaccine Intent
Description: This is the respondent's likelihood to receive the flu vaccine before the end of the flu season. This was elicited on an 11-point Likert scale (0 extremely unwilling, 10 extremely willing) after the video message treatment. We re-scaled this outcome to have a scale of 0 to 1. The reported results of the outcome compare participants in Arm A and Arm B (described in each arm/group description). For example, an intent of 0.03 indicates that participants in Arm A are 0.03 units on a scale more likely to intent to take up the flu vaccine compared to those in Arm B.
Time Frame: This outcome was assessed after the video treatment during Baseline survey, which took approximately 20 minutes.
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: units on a scale
Arm/Group | Concordant (Arm A) vs. Discordant Expert Sender (Arm B) - Black Participants | Concordant (Arm A) vs. Discordant Expert Sender (Arm B) - White Participants | Acknowledgement (Arm A) vs. Standard Signal (Arm B) - Black Participants | Layperson Sender (Arm A) vs. Expert Sender (Arm B) - Black Participants
Number analyzed (Participants) | 832 | 1221 | 827 | 845
units on a scale | .0263281 [-.0236633 to .0763195] | .0034755 [-.037638 to .044589] | .0268659 [-.0226463 to .0763781] | .0187403 [-.0305011 to .0679817]

7. Primary Outcome: COVID-19 Vaccine Intent
Description: This is the respondent's likelihood to take up the COVID-19 vaccine if made available free of charge. This was elicited on an 11-point Likert scale (0 extremely unwilling, 10 extremely willing) after the video message treatment. We re-scaled this outcome to have a scale of 0 to 1. The reported results of the outcome compare participants in Arm A and Arm B (described in each arm/group description). For example, an intent of 0.04 indicates that participants in Arm A are 0.04 units on a scale more likely to intent to take up the COVID-19 vaccine compared to those in Arm B.
Time Frame: This outcome was assessed after the video treatment during Baseline survey, which took approximately 20 minutes.
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: units on a scale
Arm/Group | Concordant (Arm A) vs. Discordant Expert Sender (Arm B) - Black Participants | Concordant (Arm A) vs. Discordant Expert Sender (Arm B) - White Participants | Acknowledgement (Arm A) vs. Standard Signal (Arm B) - Black Participants | Layperson Sender (Arm A) vs. Expert Sender (Arm B) - Black Participants
Number analyzed (Participants) | 587 | 866 | 581 | 592
units on a scale | .0350147 [-.0251663 to .0951958] | .009072 [-.0404259 to .0585699] | .0544277 [-.0064546 to .11531] | .0881949 [.0291914 to .1471983]

8. Primary Outcome: Flu Vaccine Take-up
Description: This is respondents' self-report in the follow-up survey on whether they or their family members had received the flu shot or redeemed the coupon since the intervention. The reported results of the outcome compare participants in Arm A and Arm B (described in each arm/group description). For example, 15.0 percentage points indicate that participants in Arm A are more likely to report that they and/or another household member received the flu vaccine by 15.p percentage points compared to those in Arm B.
Time Frame: This outcome was assessed during the follow-up survey which was conducted at least two weeks after the initial baseline survey.
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage points
Groups:
- Concordant (Arm A) vs. Discordant Expert Sender (Arm B) - Black Participants: This group combines the following arms to measure the effect of racial concordance between sender and receiver (i.e. intervention) among Black Participants:
  1. Black Participant-Concordant Sender-Expert Sender-Standard Signal (i.e. Arm A)
  2. Black Participant-Discordant Sender-Expert Sender-Standard Signal (i.e. Arm B)
Arm/Group | Concordant (Arm A) vs. Discordant Expert Sender (Arm B) - Black Participants | Concordant (Arm A) vs. Discordant Expert Sender (Arm B) - White Participants | Acknowledgement (Arm A) vs. Standard Signal (Arm B) - Black Participants | Layperson Sender (Arm A) vs. Expert Sender (Arm B) - Black Participants
Number analyzed (Participants) | 139 | 377 | 137 | 151
percentage points | -7.70997 [-24.9643 to 9.54435] | -01.39307 [-11.01382 to 8.22767] | -12.00413 [-28.76783 to 4.75957] | 14.96955 [-1.50779 to 31.44689]

ADVERSE EVENTS:
Time Frame: 6.5 months (3 months during the 2019 to 2020 flu season and 3.5 months during the 2020-2021 flu season)
Arm/Group | Black Participant-Concordant Sender-Expert Sender-Standard Signal | Black Participant-Concordant Sender-Lay Sender-Standard Signal | Black Participant-Discordant Sender-Expert Sender-Standard Signal | Black Participant-Discordant Sender-Expert Sender-Acknowledgement Signal | White Participant-Concordant Sender-Expert Sender-Standard Signal | White Participant-Discordant Sender-Expert Sender-Standard Signal
All-Cause Mortality (participants affected / at risk) | 0/479 | 0/496 | 0/478 | 0/485 | 0/649 | 0/658
Serious Adverse Events (participants affected / at risk) | 0/479 | 0/496 | 0/478 | 0/485 | 0/649 | 0/658
Other Adverse Events (participants affected / at risk) | 0/479 | 0/496 | 0/478 | 0/485 | 0/649 | 0/658

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-12): https://cdn.clinicaltrials.gov/large-docs/75/NCT04160975/Prot_SAP_000.pdf